CLINICAL TRIAL: NCT05672368
Title: Phase II Study of the Da Vinci Single Port (SP) Robotic System for Abdominal and Pelvic Procedures
Brief Title: The da Vinci Single Port Robotic System for Use in Abdominal and Pelvic Surgical Procedures
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 22446; NCI-2022-10346 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22446 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Disease or Disorder
MeSH Terms: conditions — Disease | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Device feasibility (da Vinci SP1098 robotic system) (Experimental): Patients undergo surgery using the da Vinci SP1098 robotic system on study.
  Interventions: Device: Robot-Assisted Surgery

INTERVENTIONS:
Device: Robot-Assisted Surgery — Undergo surgery using the da Vinci SP device
  Other Names: Navigation and Robotics; Robot Assisted; Robotic Surgery

SUMMARY:
This phase II trial test the effectiveness and safety of a single-port robotic device (the da Vinci single port [SP]1098) for use in abdominal and pelvic surgeries. The da Vinci SP1098 robotic device can be used to perform less invasive surgeries that allow entry into the body through a single, small incision. The use of this device during surgery may allow surgeons to perform complex procedures that result in less pain, fewer complications and side effects, and improved recovery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the effectiveness and safety for abdominal and pelvic procedures of a single-port robotic device (da Vinci SP1098) that is Food and Drug Administration (FDA)-approved for other indications, specifically urological and transoral otolaryngology surgical procedures.

OUTLINE:

Patients undergo surgery using the da Vinci SP1098 robotic system on study.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Any patient scheduled to undergo robot-assisted abdominal or pelvic procedures
* Age > 18 years

Exclusion Criteria:

* Body mass index (BMI) > 45
* Contraindications to minimally invasive surgery including chronic obstructive pulmonary disorders
* Past history of failed attempt of minimally invasive abdominal or pelvic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2026-01-27 (Estimated); Study Completion 2026-01-27 (Estimated)

PRIMARY OUTCOMES:
Conversion of operation to laparotomy | Within 30 days of operation
  The number and frequency will be reported with 95% confidence intervals.
Incidence of major surgical complications | Within 30 days of operation
  Will be assessed by Clavien-Dindo classification as grade 3 or higher. The number and frequency will be reported with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Moslemi-Kebria, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States